CLINICAL TRIAL: NCT03005015
Title: A Randomized Phase II Study of Lenvatinib Versus Doxorubicin in Second Line Advanced or Recurrent Endometrial Carcinoma
Brief Title: Lenvatinib in Second Line Endometrial Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: supporting company (Eisai) withdrew their interest
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1528
Record Dates: First submitted 2016-08-18; First posted 2016-12-29 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Endometrial Neoplasms
MeSH Terms: conditions — Endometrial Neoplasms | interventions — lenvatinib; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lenvatinib (Experimental): Lenvatinib 24 mg orally every day. Treatment is continued until unacceptable toxicity, progressive disease or patient withdrawal
  Interventions: Drug: Lenvatinib
- Doxorubicin (Active Comparator): Doxorubicin 60 mg/m² iv bolus every 3 weeks. Treatment is continued for a maximum of 6 cycles or until unacceptable toxicity, progressive disease or patient withdrawal.
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Drug: Lenvatinib
  Arms: Lenvatinib
Drug: Doxorubicin
  Arms: Doxorubicin

SUMMARY:
The primary objective of this multicenter, randomized phase II trial is to assess the efficacy, as measured by progression-free survival (PFS), of lenvatinib compared to doxorubicin in advanced or recurrent endometrial cancer.

The main secondary objective is to evaluate the predictive value of Ang-2 on lenvatinib activity and establishing a cutoff value as potential selection criteria for phase III.

Other secondary objectives are to assess the tolerability and safety of lenvatinib in this setting and overall survival, response and disease control.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects age ≥18 years at the time of informed consent
* World Health Organization (WHO) Performance Status of 0 or 1
* Patients with histologically confirmed endometrial cancer including serous-papillary and clear cell histologies. Uterine carcinosarcomas are allowed.
* Radiographic evidence of disease progression according to RECIST 1.1 after 1 prior systemic, platinum-based chemotherapy regimen for metastatic or primary unresectable endometrial carcinoma for which no surgical or radiotherapy treatment options exist.
* Patients with disease progression following platinum-based chemotherapy administered as either adjuvant or neoadjuvant treatment are also eligible.
* Patients may have received prior radiotherapy and / or adjuvant chemotherapy for early high-risk disease
* Patients may not have received prior treatment with anthracyclines
* Blood samples available for retrospective central assessment of Ang-2 level
* Patients may have had prior therapy providing the following conditions are met:
* Surgery and radiation therapy: wash-out period of 14 days and subjects must have recovered adequately from any toxicity and/or complications from radiotherapy and major surgery prior to starting therapy.
* Systemic anti-tumor therapy or any investigational agent: wash-out period of 21 days (or 5 x half-life)
* Recovery from any toxic effects of prior therapy to ≤ Grade 1 per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v4.) except alopecia
* Adequate contraceptive measures
* Signed written informed consent

Exclusion Criteria:

* Inadequate hematologic, renal and hepatic functions
* Abnormal cardiac function

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 2.5 years
  PFS assessed by Response Evaluation Criteria in Solid Tumors (RECIST

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Casado, Study Chair — Hospital Universitario San Carlos, Madrid, Spain
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland